CLINICAL TRIAL: NCT07339384
Title: Circulating Tumor DNA Assessment in Early-Stage Endometrial Cancer (SIGNAL-EMC 101)
Brief Title: Signatera Assessment in Early-Stage Endometrial Cancer
Acronym: SIGNAL-EMC 101
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-102-NCP
Record Dates: First submitted 2025-12-30; First posted 2026-01-14 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer
Keywords: ctDNA; Endometrial Cancer; circulating tumor; Signatera; Molecular Residual Disease; MRD; biomarker-guided therapy; Vaginal Brachytherapy; VBT; High-Intermediate Risk Endometrial Cancer; Adjuvant Therapy; Tumor-informed assay
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Following the initial baseline test, providers in Arm A will be blinded to all subsequent ctDNA results unless ctDNA positive within the first 12 weeks in Arm A (in which case, the provider will be notified and TPC will be initiated).
  Providers treating participants in Arm B will remain blinded to all ctDNA results following the initial baseline test. Providers and patients enrolled in the early stage low-risk and high-risk cohorts will be blinded to all ctDNA results (post-operatively, during treatment, and during surveillance).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Observation (Other): Participants will be monitored by their study physician and will not receive treatment
  Interventions: Device: Signatera Genome ultra-sensitive ctDNA blood test
- Vaginal Brachytherapy (VBT) (Active Comparator): Participants will receive standard-of-care vaginal brachytherapy
  Interventions: Device: Signatera Genome ultra-sensitive ctDNA blood test

INTERVENTIONS:
Device: Signatera Genome ultra-sensitive ctDNA blood test — Signatera Genome is intended for use as a post-surgical risk stratification tool for patients with early-stage HIR endometrial cancer. The test is used to identify patients with no evidence of MRD following definitive surgery.

SUMMARY:
The goal of this clinical trial is to assess if circulating tumor DNA can guide adjuvant selection in high-intermediate risk early-stage endometrial cancer. The main question it aims to answer is:

• To evaluate if 3-year recurrence-free survival among women with Stage I, high-intermediate risk endometrial cancer who are ctDNA negative after receiving ctDNA-guided observation is non-inferior to adjuvant vaginal brachytherapy (an internal radiation therapy) Researchers will compare high-risk intermediate ctDNA negative participants who are observed to those who receive vaginal brachytherapy to see if they have similar outcomes.

Participants will be asked to:

* Receive serial ctDNA testing
* Visit their study doctor per their standard of care visits about every 3 months for 2 years
* Answer a questionnaire about their well-being

DETAILED DESCRIPTION:
This includes a randomized, multi-center, non-inferiority trial for a biomarker-defined subgroup, alongside two parallel, non-randomized exploratory cohorts. The study utilizes a biomarker-stratified design to formally test a treatment de-escalation strategy in patients with HIR endometrial cancer.

Following surgery, patients in the HIR cohort will be stratified based on post-operative circulating tumor DNA (ctDNA) status, as determined by the Signatera Genome assay. ctDNA-negative HIR Patients, based on the first valid post-operative ctDNA result within the baseline window, will be randomized (1:1) to either:

* Arm A: Observation unless ctDNA positivity within baseline window (<12 weeks), with serial ctDNA monitoring.
* Arm B: Vaginal brachytherapy (VBT) with serial ctDNA monitoring.

Following the initial baseline test, providers will be blinded to subsequent ctDNA results unless ctDNA positive within the first 12 weeks in Arm A [in which case, the provider will be notified and treatment of physician's choice (TPC) will be initiated. Initiation of TPC following ctDNA conversion is considered part of the ctDNA-guided treatment strategy, not a protocol deviation or cross-over, and such patients remain in the intent-to-treat population in Arm A]. Providers treating patients in Arm B will remain blinded to all ctDNA results after randomization. Post-operative ctDNA-Positive HIR patients will not be randomized and will continue serial testing while receiving TPC, which may include observation, radiation and/or chemotherapy. Providers and patients will be unblinded to the initial ctDNA result and blinded to ctDNA results thereafter.

The study will also include early stage low-risk (LR) and high-risk (HR) cohorts. Patients in these cohorts will not be randomized. They will continue serial ctDNA testing while receiving TPC, which may include observation, radiation and/or chemotherapy, and during surveillance. Providers and patients will be blinded to ctDNA results during the post-operative, TPC and surveillance period.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria includes the following selection criteria to be eligible for inclusion in any aspect of the study. Eligibility will be assessed by the investigator:

1. Signed and dated informed consent form (ICF) obtained prior to any trial-specific enrollment procedure.

2. Patient is ≥ 18 years-old at the time of ICF signature. 3. Able to submit sufficient residual tissue obtained per standard of care procedures.

HIR patients must meet all the following selection criteria to be eligible for the randomization cohort in the study. Eligibility will be assessed by the investigator:

1. FIGO 2009 Stage I after hysterectomy and lymph node assessment by bilateral pelvic lymphadenectomy or SLND

   1. If para-aortic lymph nodes are not pathologically assessed, documentation of surgical assessment or imaging is recommended.
2. Stage I patients with endometrioid histology:

   1. Age 70 years or older with one uterine risk factor,
   2. Age 50-69 years with two risk factors,
   3. Age 18 - 49 years with three risk factors.

Uterine risk factors include:

* Grade 2 or 3 tumor.
* Outer half depth of invasion.
* Lymphovascular invasion. Note: peritoneal cytology must be negative if performed.

Patients must meet all the following selection criteria to be eligible for the observation arms of the study. Eligibility will be assessed by the investigator following hysterectomy and lymph node assessment by bilateral pelvic and para-aortic lymphadenectomy or SLND:

1. High risk cohort

a. FIGO 2009 Stage I with high risk histology i. Defined as serous, clear cell, carcinosarcoma, or mixed histology.

1. Negative peritoneal cytology, where performed (recommended)
2. If para-aortic lymph nodes are not pathologically assessed, imaging is required b. FIGO 2009 Stage II Endometrioid

2. Low risk cohort

a. FIGO 2009 Stage I patients at low risk of recurrence i. Endometriod histology ii. Absent uterine risk factors, or present but insufficient to meet HIR criteria

Exclusion Criteria:

Patients are not eligible for the study if they meet any of the following criteria, as assessed by the investigator:

1. Undifferentiated or dedifferentiated histology
2. Uterine sarcoma
3. Prior pelvic radiation therapy
4. Positive pelvic washings
5. Pelvic lymph node assessment was not performed
6. Isolated Tumor Cells (ITC) identified in the lymph node(s)
7. Prior therapy for endometrial cancer (including hormonal therapy, chemotherapy, targeted therapy, immunotherapy)

   a. Contraceptives or other hormonal management for endometrial intraepithelial hyperplasia is allowed
8. Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of active malignancy within the last five years.

   a. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy.
9. Patients with a history of serious comorbid illness or uncontrolled illnesses that would preclude protocol therapy.
10. Patients with a history of myocardial infarction, unstable angina, or uncontrolled arrhythmia within 3 months from enrollment.
11. Previous diagnosis of Crohn's disease or ulcerative colitis.
12. Patient is currently receiving, or plans to receive, commercial ctDNA/MRD assay for disease monitoring, excluding Signatera. Patients must agree to forego testing with assays other than Signatera Genome upon enrollment until end of study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1010 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2034-05 (Estimated); Study Completion 2034-05 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival (RFS) | 3 years from randomization to the first occurrence of disease recurrence or death from any cause, whichever occurs first
  The primary objective of this study is to evaluate if recurrence free survival (RFS) is non-inferior among women with stage I high-intermediate risk endometrial cancer who are ctDNA-negative after surgery and managed with ctDNA-guided observation versus adjuvant VBT.

SECONDARY OUTCOMES:
Overall Survial | From enrollment to Year 3 and enrollment to Year 5
  Comparison of overall survival (OS) among all high-intermediate risk (HIR) patients and recurrence free survival (RFS) across treatment groups and assess whether ctDNA-guided de-escalation group is non-inferior to adjuvant VBT.
ctDNA Clearance Rate | From enrollment until first surveillance visit at 12 weeks
  Estimate the ctDNA clearance rate among high-intermediate risk ctDNA positive participants.
Clinicopathologic and Molecular Risk Factors | Up to 5 years from enrollment
  Assess the primary and secondary objectives by clinicopathologic and molecular (e.g. POLE, MMR-D, p53 aberrant, p53 wild type) risk factors, and ethnic/racial groups among high-intermediate risk patients.

OTHER OUTCOMES:
Lead time of ctDNA positivity | Up to 5 years from enrollment
  Examine differences in lead time of ctDNA positivity relative to clinical or radiologic diagnosis of recurrence across different ctDNA dynamic groups (e.g. clearance, persistent negative) among LR, HIR, and HR patients.
Disease-specific recurrence | At 3 years and 5 years.
  Determine disease-specific recurrence among high-intermediate risk patients.
ctDNA positivity rate | From randomization to 3 years and 5 years
  Assess ctDNA positivity rate, defined as proportion of patients, among all HIR, HR, and LR patients with evaluable ctDNA results
ctDNA negativity rate | From randomization to 3 years and 5 years
  ctDNA negativity rate, defined as proportion of patients with a negative ctDNA, among all HIR, HR, and LR patients with evaluable ctDNA results.
ctDNA clearance rate | From enrollment up to 5 years
  Assess the ctDNA clearance rate of ctDNA from HIR, HR, and LR participants.
ctDNA negative persistence rate | From enrollment to end of treatment and up to 5 years.
  Assess proportion of HIR, HR, and LR participants who remain ctDNA-negative throughout the surveillance period among participants who were ctDNA-negative post-operatively or post-adjuvant treatment.
Mean Tumor Molecules (MTM) | From enrollment to up to 5 years
  Assess mean tumor molecules (MTM) presence change over time in HIR, HR, and LR participants.
Variant Allele Frequencies (VAF) | From enrollment up to 5 years
  Assess variant allele frequencies (VAF) changes over time in HIR, HR, and LR participants.
Cost-effectiveness of ctDNA guided care | Up to 5 years from enrollment
  Compare the ctDNA cost for High-Risk Intermediate endometrial cancer participants who were randomized to the observation cohort to those that received standard of care (VBT) treatment
Quality of Life Outcomes | Up to 5 years from enrollment
  Compare Quality of Life (QoL) outcomes between the Observation and Vaginal Brachytherapy (VBT) treatment arms among HIR patients, utilizing the Functional Assessment of Cancer Therapy - Endocrine Symptoms Version 4 (FACT-ES) patient-reported outcome (PRO).

CONTACTS AND LOCATIONS:
Overall Officials: Adam ElNaggar, MD, Study Director — Natera, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Firth, D. (1993). Bias reduction of maximum likelihood estimates. Biometrika, 80(1), 27-38
- [Background] Mahdi H, Elshaikh MA, DeBenardo R, Munkarah A, Isrow D, Singh S, Waggoner S, Ali-Fehmi R, Morris RT, Harding J, Moslemi-Kebria M. Impact of adjuvant chemotherapy and pelvic radiation on pattern of recurrence and outcome in stage I non-invasive uterine papillary serous carcinoma. A multi-institution study. Gynecol Oncol. 2015 May;137(2):239-44. doi: 10.1016/j.ygyno.2015.01.544. Epub 2015 Jan 29. PMID 25641568
- [Background] Creutzberg CL, van Putten WL, Warlam-Rodenhuis CC, van den Bergh AC, de Winter KA, Koper PC, Lybeert ML, Slot A, Lutgens LC, Stenfert Kroese MC, Beerman H, van Lent M; postoperative Radiation Therapy in Endometrial Carcinoma Trial. Outcome of high-risk stage IC, grade 3, compared with stage I endometrial carcinoma patients: the Postoperative Radiation Therapy in Endometrial Carcinoma Trial. J Clin Oncol. 2004 Apr 1;22(7):1234-41. doi: 10.1200/JCO.2004.08.159. PMID 15051771
- [Background] Proceedings of the International Conference on the Haemophilus, Actinobacillus and Pasteurella (HAP) Group of Organisms. June 1989. Can J Vet Res. 1990 Apr;54 Suppl:S1-82. No abstract available. PMID 2361201
- [Background] Siegenthaler F, Lindemann K, Epstein E, Rau TT, Nastic D, Ghaderi M, Rydberg F, Mueller MD, Carlson J, Imboden S. Time to first recurrence, pattern of recurrence, and survival after recurrence in endometrial cancer according to the molecular classification. Gynecol Oncol. 2022 May;165(2):230-238. doi: 10.1016/j.ygyno.2022.02.024. Epub 2022 Mar 8. PMID 35277281
- [Background] Lund L, Christiansen UB, Hansen IM, Funder VT. Carcinoma presenting as intrarenal haematoma, either spontaneously or after minor trauma. Int Urol Nephrol. 1994;26(5):497-500. doi: 10.1007/BF02767648. PMID 7860194
- [Background] Adib SM, Hajjar H, Lawand T. Cost and length-of-stay of hospital care billed to the Ministry of Public Health by private hospitals. J Med Liban. 1997;45(1):4-9. PMID 9421940
- [Background] Kemppainen TA, Kosma VM, Janatuinen EK, Julkunen RJ, Pikkarainen PH, Uusitupa MI. Nutritional status of newly diagnosed celiac disease patients before and after the institution of a celiac disease diet--association with the grade of mucosal villous atrophy. Am J Clin Nutr. 1998 Mar;67(3):482-7. doi: 10.1093/ajcn/67.3.482. PMID 9497194
- [Background] Curti HJ, Sanches PC, Jabur Filho M, Mazzoni CJ, Pasian S, Carvalhal SS. [Sudden death in a low socioeconomic population of the city of Campinas: anatomopathological study]. Arq Bras Cardiol. 1983 Aug;41(2):109-14. No abstract available. Portuguese. PMID 6675596
- [Background] Miteva L, Mitev V, Durmishev A. [The role of a growth-related cytosol protein kinase in the pathogenesis of psoriasis]. Eksp Med Morfol. 1994;32(3-4):19-26. Bulgarian. PMID 8857029
- [Background] https://seer.cancer.gov/csr/1975_2018/
- [Background] Sohaib SA, Houghton SL, Meroni R, Rockall AG, Blake P, Reznek RH. Recurrent endometrial cancer: patterns of recurrent disease and assessment of prognosis. Clin Radiol. 2007 Jan;62(1):28-34; discussion 35-6. doi: 10.1016/j.crad.2006.06.015. PMID 17145260
- [Background] Howlader N, N.A., Krapcho M, Miller D, Brest A, Yu M, Ruhl J, Tatalovich Z, Mariotto A, Lewis DR, Chen HS, Feuer EJ, Cronin KA (eds), SEER Cancer Statistics Review, 1975-2017. National Cancer Institute. Bethesda, MD
- [Background] Siegel RL, Kratzer TB, Giaquinto AN, Sung H, Jemal A. Cancer statistics, 2025. CA Cancer J Clin. 2025 Jan-Feb;75(1):10-45. doi: 10.3322/caac.21871. Epub 2025 Jan 16. PMID 39817679
- [Background] van den Heerik ASVM, Horeweg N, Creutzberg CL, Nout RA. Vaginal brachytherapy management of stage I and II endometrial cancer. Int J Gynecol Cancer. 2022 Mar;32(3):304-310. doi: 10.1136/ijgc-2021-002493. PMID 35256416
- [Background] Kako TD, Kamal MZ, Dholakia J, Scalise CB, Arend RC. High-intermediate risk endometrial cancer: moving toward a molecularly based risk assessment profile. Int J Clin Oncol. 2022 Feb;27(2):323-331. doi: 10.1007/s10147-021-02089-2. Epub 2022 Jan 17. PMID 35038071